CLINICAL TRIAL: NCT05073185
Title: Characterizing Resilience to Food-cue Induced Overeating in Children
Brief Title: Resilience to the Effects of Advertising in Children
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: University of Kansas Medical Center (Other); University of Missouri, Kansas City (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Professor, Penn State University
Other Study IDs: Project REACH; R01DK126050 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-10-11 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Childhood
Keywords: Obesity; food-cue reactivity; functional magnetic resonance imaging; eating behaviors; food marketing; food advertisement
MeSH Terms: conditions — Pediatric Obesity; Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with healthy weight status: 100 child-parent dyads (200 total) will be followed for 1 year to determine the behavioral and neural impact of food and toy advertising exposure. Children will be 7-9 years old, with body mass index < 85th % for age and sex, and either with a mother who has BMI of 30 kg/m-sq or over or a BMI of 25 kg/m-sq or less.

SUMMARY:
Strong empirical evidence shows food marketing promotes excess energy intake and obesity. Yet, not all children are susceptible to its effects and this variability is poorly understood. Identifying sources of this variability is a public health priority not only because it may elucidate characteristics of children who are most susceptible, but also because it may highlight novel sources of resiliency to overconsumption. The proposed research will use state-of-the art, data-driven approaches to identify neural, cognitive and behavioral phenotypes associated with resiliency to food-cue (i.e. food advertisement) induced overeating and determine whether these phenotypes protect children from weight gain during the critical pre-adolescent period.

DETAILED DESCRIPTION:
The investigator's central hypothesis is that children who are resistant to food-cue induced overeating will exhibit a distinct cluster of neural, behavioral, and cognitive traits that protect them from weight gain, even in the context of high-familial obesity risk. Identifying these traits is critical to the development of successful, individually tailored obesity prevention programs. This hypothesis is informed by compelling preliminary research showing that children who are less susceptible to food-cue induced eating in the laboratory show decreased neural activation in somatosensory (i.e., post-central gyrus) and reward (i.e., striatum) regions and increased activation in cognitive control regions (i.e., dorsolateral prefrontal cortex-dlPFC) following food commercial exposure.

These results provide a strong foundation for characterizing neural responses that are associated with resiliency to food-cue induced eating, but highlight major gaps in the literature that must be addressed to advance the field. This proposal will make three novel contributions to the understanding of the etiology of obesity. Using a prospective, family-risk design, the investigators will follow 100, 7-9 year-old children who have healthy weight but vary by risk for obesity (based on maternal weight status) for 1 year to characterize neural and behavioral responses to food commercials and identify common neural networks associated with resiliency to food-cue induced overconsumption. Second, the investigators will use sophisticated behavioral coding to characterize children's eating following food commercial exposure at both homeostatic (i.e., meal consumed when hungry) and non-homeostatic (i.e., eating in the absence of hunger - EAH snack buffet) events and relate individual differences in eating behavior to neural phenotypes. Finally, the investigators will follow children over 1 year to determine whether the neural and behavioral responses at baseline are protective against adiposity gains, during a critical period where children are cognizant of the purpose of advertising, but cannot fully defend against its effects.

Baseline data will be collected over 4 weekly initial visits, followed by a 5th visit one year later.

ELIGIBILITY:
Child Inclusion Criteria:

1. In order to be enrolled, children must be of good health based on parental self-report.
2. Have no learning disabilities (e.g., ADHD).
3. Have no allergies to the foods or ingredients used in the study.
4. Not be claustrophobic.
5. Not be taking any medications known to influence body weight, taste, food intake, behavior, or blood flow.
6. Be 7-9 years-old at enrollment.
7. The child must speak English.

Parent Inclusion Criteria:

1. The parent who has the most knowledge of the child's eating behavior, media access, sleep and behavior must be available to attend the visits with their child. This would be decided among the parents.
2. The biological mother must have a body mass index either between 18.5 - 25 kg/m2 (low-risk group) or greater than or equal to 30 kg/m2 (high-risk group). One parent can report on both parents' BW and height.

Exclusion Criteria:

Children would be excluded if:

1. They are not within the age requirements (< than 7 years old or > than 9 years-old at baseline).
2. If they are taking cold or allergy medication, or other medications known to influence cognitive function, taste, appetite, or blood flow.
3. If they don't speak English.
4. If they are colorblind
5. If they report being claustrophobic.
6. if they have a learning disability, ADD/ADHD, language delays, autism or other neurological or psychological conditions.
7. if they have a pre-existing medical condition such as type I or type II diabetes, rheumatoid arthritis, Cushing's syndrome, Down's syndrome, food allergies, severe lactose intolerance, Prader-Willi syndrome, HIV, cancer, renal failure, or cerebral palsy.
8. if they are allergic to foods or ingredients used in the study.
9. if they have tattoos, permanent makeup, dental ware, pacemakers, or metal implants that would preclude safe completion of the MRI.
10. if the child has had an X-ray in the month prior to Visits 1 and 6. If so, they will be scheduled at a later date.

Parent Exclusion Criteria:

1. if the biological mother has a body mass index < 18.5 kg/m2
2. if the mother is between 25-30 kg/m2.
3. if the parent is unable to attend the study visits
4. if the family reports plans to move away from the area in the next year.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents and children meeting the eligibility criteria living within 40 miles of University Park, Pa.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
fMRI blood oxygen level dependent (BOLD) response to food commercials | baseline
  Whole-brain response to food commercials, followed by images of high and low energy density foods in a fMRI scan
fMRI blood oxygen level dependent (BOLD) response to toy commercials | baseline
  Whole-brain response to toy commercials, followed by images of high and low energy density foods in a fMRI scan
Food intake in grams after no commercial viewing | baseline
  Intake in grams from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in kcals after no commercial viewing | baseline
  Intake in kcals from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in grams after viewing food commercials | baseline
  Intake in grams from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in kcals after viewing food commercials | baseline
  Intake in kcals from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in grams after food commercial viewing | 1 year
  Intake in grams from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in kcals after food commercial viewing | 1 year
  Intake in kcals from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in grams after viewing toy commercials | baseline
  Intake in grams from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Food intake in kcals after viewing toy commercials | baseline
  Intake in kcals from an eating in the absence of hunger paradigm consumed following advertisement exposure when children are not hungry (i.e., non-homeostatic intake)
Video recording of meal and EAH snack buffet | baseline
  A digital recording of the Child eating the Test Meal and the EAH snack buffet will be saved. We have developed a behavior coding technique to count specific behaviors while the child eats. We will also be transcribing the audio.
Video recording of meal and EAH snack buffet | 1 year
  A digital recording of the Child eating the Test Meal and the EAH snack buffet will be saved. We have developed a behavior coding technique to count specific behaviors while the child eats. We will also be transcribing the audio.
Change from baseline DXA analysis for total body fat mass of child at 1 year | baseline
  Examine change in children's fat mass index = total fat mass(kg) / height (m2)
fMRI Region of Interest (ROI) response to toy commercials and subsequent views of high and low energy density food pictures. | baseline
  We will examine the strength of the neural connections between reward/somatosensory and cognitive control regions.
fMRI Region of Interest (ROI) response to food commercials and subsequent views of high and low energy density food pictures. | baseline
  We will examine the strength of the neural connections between reward/somatosensory and cognitive control regions.

SECONDARY OUTCOMES:
Change in Android fat mass as measured by DXA analysis | Baseline and 1 year
  Android fat mass (%) = (Android fat mass (kg) / total fat mass (kg))*100
Change in Gynoid fat mass as measured by DXA analysis | Baseline and 1 year
  Gynoid fat mass (%) = (Gynoid fat mass (kg) / total fat mass (kg))*100
Child screen time | Baseline and 1 year
  Child questionnaire quantifying the number of hours per day a child is exposed to different types of media.
Child's brand awareness | Baseline and 1 year
  Child's brand awareness assessed by a child computerized task. Children are asked to match pictures of products and brand logos. No scaling is used.
Change in scores from the NIH Toolbox: Child Cognitive battery-Flanker test | Baseline and 1 year
  The Flanker is a measure of executive function, specifically tapping inhibitory control and attention. Scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these "vectors" ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value from 0-10. For any given individual, accuracy is considered first. If accuracy levels for the participant are less than or equal to 80%, the final "total" computed score is equal to the accuracy score. If accuracy levels for the participant reach more than 80%, the reaction time score and accuracy score are combined. Higher scores indicate higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli.
Change in scores from the NIH Toolbox: Child Cognitive battery-List Sorting Working memory test | Baseline and 1 year
  The List Sorting Working memory test assesses working memory. The List Sorting test requires immediate recall and sequencing of different visually and orally presented stimuli (i.e., "working memory"). Pictures of different foods and animals are displayed with accompanying audio recording and written text (e.g., "elephant"), and the participant is asked to say the items back in size order from smallest to largest, first within a single dimension (either animals or foods, called 1-List) and then on two dimensions (foods, then animals, called 2-List). The test takes approximately seven minutes to administer. List Sorting is scored by summing the total number of items correctly recalled and sequenced on 1-List and 2-List, which can range from 0-26.Higher scores on each of these indicate higher levels of working memory within the normative standard being applied.
Change in scores from the NIH Toolbox: Child Cognitive battery-Dimensional Change Card Sort Test (DCCS) | Baseline and 1 year
  The Dimensional Change Card Sort Test is used to measure cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, scores ranging from 0-10. For any given individual, accuracy is considered first. If accuracy levels for the participant are less than or equal to 80%, the final "total" computed score is equal to the accuracy score. If accuracy levels for the participant reach more than 80%, the reaction time score and accuracy score are combined. Higher scores indicate higher levels of cognitive flexibility.

OTHER OUTCOMES:
Height of child and one parent | Baseline
  Height (cm) will be measured. Body mass index (BMI) and BMI z scores will be calculated.
Weight of child and one parent | Baseline
  Weight (kg) will be measured. Body mass index (BMI) and BMI z scores will be calculated.
Height of child and one parent | 1 year
  Height (cm) will be measured. Body mass index (BMI) and BMI z scores will be calculated.
Weight of child and one parent | 1 year
  Weight (kg) will be measured. Body mass index (BMI) and BMI z scores will be calculated.
Taste testing to measure liking of foods | Baseline
  Ratings of how much a child likes a food is measured on a computerized visual scale. The scale is from 1 (Hate It) to 5 (Love It).
Taste testing to measure liking of foods | 1 Year
  Ratings of how much a child likes a food is measured on a computerized visual scale. The scale is from 1 (Hate It) to 5 (Love It).
IQ test results | Baseline
  The child will be given an IQ test (Wechsler Abbreviated Scale of Intelligence) to determine cognitive ability measures. It is a battery of two subtests: Vocabulary (31-item) and Matrix Reasoning (30-item). Each of the 2 subtests is scored by taking a sum of all items and referencing and age- and sex-normed tables to get standardized scores; these standardized scores are then added to get the 3 subscale scores, their associated IQ scores percentiles; Higher scores indicate a higher IQ.
IQ test results | 1 year
  The child will be given an IQ test (Wechsler Abbreviated Scale of Intelligence) to determine cognitive ability measures. The WASI is a battery of two subtests: Vocabulary (31-item) and Matrix Reasoning (30-item). Each of the 2 subtests is scored by taking a sum of all items and referencing and age- and sex-normed tables to get standardized scores; these standardized scores are then added to get the 3 subscale scores, their associated IQ scores percentiles; Higher scores indicate a higher IQ.
Freddy Fullness survey | Baseline
  Child fullness will be measured using a pictorial fullness scale termed a Freddy Fullness scale. Prior to the visit, children will be instructed to fast for at least 3hrs. They are then instructed on use of the scale by trained research personnel. Following this, children will be asked to report current fullness on the scale, which measures a fullness range of 0 to 150 mm. They will be asked to make a total of 2 ratings using this scale, one immediately before each meal, and one following the meal.
Freddy Fullness survey | 1 year
  Child fullness will be measured using a pictorial fullness scale termed a Freddy Fullness scale. Prior to the visit, children will be instructed to fast for at least 3hrs. They are then instructed on use of the scale by trained research personnel. Following this, children will be asked to report current fullness on the scale, which measures a fullness range of 0 to 150 mm. They will be asked to make a total of 2 ratings using this scale, one immediately before each meal, and one following the meal.
Physical Activity Intensity | Baseline
  An ActiGraph watch will be given to the parent with instruction. The child will be wearing the wrist watch for one week in the baseline time period (other than when showering, bathing or in a pool) and will hand it back at their next visit.
Sleep Quality and Sleep Quantity | Baseline
  An ActiGraph watch will be given to the parent with instruction. The child will be wearing the wrist watch for one week in the baseline time period (other than when showering, bathing or in a pool).
Computer game called Stop Signal Task | Baseline
  The stop signal task (SST) is used to capture individual differences in response inhibition. There is no max/min range for performance. For both the Stop-signal reaction time and the stop-signal delay: lower values indicate better control. This is administered in the fMRI scanner.
Television and internet use and exposure assessment | Baseline
  Parent reported questionnaires of television and internet use and exposure to shows and commercials
Television and internet use and exposure assessment | 1 year
  Parent reported questionnaires of television and internet use and exposure to shows and commercials
Child pubertal development assessment | Baseline
  Parental questionnaire:Child Puberty and Tanner Questionnaire. Scoring: Male genitals are scored on a scale of 1 to 5 maturity, female breasts on a scale of 1 to 5 and both males and females on a scale of 1 to 5 for pubic hair quality and extension. Higher values indicate more pubertal development.
Child pubertal development assessment | 1 year
  Parental questionnaire:Child Puberty and Tanner Questionnaire. Scoring: Male genitals are scored on a scale of 1 to 5 maturity, female breasts on a scale of 1 to 5 and both males and females on a scale of 1 to 5 for pubic hair quality and extension. Higher values indicate more pubertal development.
Parental feeding strategies assessment | Baseline
  Parental questionnaire: Child Feeding Questionnaire (CFQ). Scored on a scale of 1-5 with lower values being better (score is the average of items for each subscale).
Child eating behavior assessment | Baseline
  Parental questionnaire: The Child Eating Behaviour Questionnaire (CEBQ) was designed to assess children's eating scale styles. It is a parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. It is made up of eight scales: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness.
Child Eating Assessment | 1 Year
  Parent Questionnaire: Parental questionnaire: The Child Eating Behavior Questionnaire (CEBQ) was designed to assess children's eating scale styles. It is a parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. It is made up of eight scales: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness.
Behavioral avoidance/inhibition assessment | Baseline
  Behavioral Avoidance/Inhibition Scale Questionnaire. The BIS/BAS Scale is a self-report questionnaire designed to measure two motivational systems: the behavioral inhibition system (BIS), which corresponds to motivation to avoid aversive outcomes, and the behavioral activation system (BAS), which corresponds to motivation to approach goal-oriented outcomes. Participants respond to questions using a 4-point Likert scale. The scale has four subscales; BAS Drive, BAS Fun Seeking, BAS Reward Responsiveness and BIS. Higher values suggest more drive, increased fun seeking, responsiveness to reward, and avoidance of unpleasantness.
Child behavior assessment | Baseline
  Parental questionnaire: The Child Behavior questionnaire (CBQ) is an assessment of temperament.Children are assessed on 15 primary temperament characteristics using a 7 point Likert scale.
Child behavior assessment | 1 Year
  Parental questionnaire: The Child Behavior questionnaire (CBQ) is an assessment of temperament.Children are assessed on 15 primary temperament characteristics using a 7 point Likert scale.
Assessment of child leisure activities | Baseline
  Parental questionnaire; Children's Leisure Activities Study Scale (CLASS). This questionnaire asks how much time the child spends in numerous types of physical activity. It is a count of time spent, not a scale.
Assessment of child leisure activities | 1 Year
  Parental questionnaire; Children's Leisure Activities Study Scale (CLASS). This questionnaire asks how much time the child spends in numerous types of physical activity. It is a count of time spent, not a scale.
Child sleep assessment | Baseline
  Parental questionnaire: Child sleep questionnaire contains 8 questions describing a child's sleep habits. The answers are on a 3 point scale with an opportunity to note if the answer indicates a problem.
Child sleep assessment | 1 Year
  Parental questionnaire: Child sleep questionnaire contains 8 questions describing a child's sleep habits. The answers are on a 3 point scale with an opportunity to note if the answer indicates a problem.
External food cue responsiveness assessment | Baseline
  Parental questionnaire: External Food Cue Responsiveness Scale Questionnaire. Nine questions are asked related to external food cues, answered in a 1 (never) -5 (always) scale. Higher scores indicate an increased responsiveness to external food cues.
Parent Alcohol Use | Baseline
  Parent questionnaire:Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed to assess alcohol consumption, drinking behaviors, and alcohol-related problems. A score of 0 (nondrinker) to 40 is possible. A score of 8 or more indicates a strong likelihood of hazardous or harmful alcohol consumption.
Parent Alcohol Use | 1 year
  Parent questionnaire: Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed to assess alcohol consumption, drinking behaviors, and alcohol-related problems. A score of 0 (nondrinker) to 40 is possible. A score of 8 or more indicates a strong likelihood of hazardous or harmful alcohol consumption.
Behavior Rating Inventory of Executive Function | Baseline
  Parent questionnaire: Behavior Rating Inventory of Executive Function (BRIEF-2) assesses executive function and self-regulation. Questions are answered on a 3-point scale (never, sometimes, often). This rating is scored by taking a sum of all items and referencing and age- and sex-normalized tables to get T-scores and percentiles; Higher T-scores indicate less Executive Function.
Household Food Security Survey Module | Baseline
  Parent questionnaire: Household Food Security Survey Module (HFFSM). Households are classified into food security status categories (1) food secure (fewer than 3 food-insecure responses); (2) low food security (more than 2 but fewer than 8 food-insecure responses among households with children); and (3) very low food security (8 or more food-insecure responses among the 18 questions for households with children) based on the number of food-insecure responses to questions. The scales differ on each question, but higher overall scores correspond with greater food insecurity. Families are said to be food insecure if they fall in categories 2 or 3.
Household Food Insecurity Access Scale | Baseline
  Parent questionnaire: Household Food Insecurity Access Scale (HFIAS). The HFIAS consists of two types of related questions. The first question type is called an occurrence question. There are nine occurrence questions that ask whether a specific condition associated with the experience of food insecurity ever occurred during the previous four weeks (30 days). Each severity question is followed by a frequency-of-occurrence question, which asks how often a reported condition occurred during the previous four weeks (1 = rarely, 2 = sometimes, 3 = often). Scoring ranges from 0-27, with higher scores indicating more food insecurity.
Community Childhood Hunger ID Project | Baseline
  Parent questionnaire: Community Childhood Hunger ID Project (CCHIP) is regarded as a model for measuring hunger in low-income families. A series of 8 questions are asked about child hunger in light of available resources, with yes or no as possible answers. Children are classified into one of 3 categories. A child is "not hungry" with a score of 0 affirmatives, "at risk" with 1-4 and "hungry" with 5 or more.
Fulkerson Home Food Inventory | Baseline
  Parental questionnaire assessing the types of food kept in the home food inventory
Demographics | Baseline
  Parent questionnaire: information describing the cultural, social and financial characteristics of the family.
Demographics | 1 Year
  Parent questionnaire: information describing the cultural, social and financial characteristics of the family.
Reinforcement Learning | Baseline
  The Behavioral Choice Task (Relative Reinforcing Value Task) is a computer task developed for use of reinforcement paradigms in humans. It has the ability to measure reinforcing value of food and toys through the use of flexible reinforcement schedules.
Decision Making in Children | Baseline
  Modified version of a decision-making task developed by Kool et al. (2017), which examine model-based decision making via the manipulation of high and low stake rewards.
Personality Traits in Children | Baseline
  Child questionnaire: alternative design to the Big Five Model, used to measure personality traits using images. There are 15 items (3 items from each scale: extraversion, neuroticism, openness, agreeableness, and conscientiousness), which are answered on a 3-point scale.
Stress in Children | Baseline
  Child questionnaire: 21 item questionnaire developed to assess stress (physical and emotional) in children. The questions are answered using a 4-point Likert scale (1=never, 4 = very often).
Loss of Control Eating in Children | Baseline
  Child questionnaire: the questionnaire assesses whether someone experienced a subjective episode of loss of control eating in the past three months. If answered "Yes", participants are instructed to respond to additional questions on before, during and after the loss of control eating occurred. No scaling is used.
Perceived Stress Scale | Baseline
  Parent questionnaire: The Perceived Stress Scale (PSS) is used to understand how different situations affect our perceived stress. The questions ask about feelings and thoughts over the past 3 months. Questions are answered using 5 points (0 = never, 4 = very often) Likert scale. 4 questions are reversed scored (0 = 4, 4 = 0). Scores from 0-13 indicate low stress, 14-26 indicate moderate stress, 27-40 indicate high stress.
Confusion, Hubbub and Order Scale | Baseline
  Parent questionnaire: Confusion, Hubbub and Order Scale (CHAOS) is a 15 question survey describing the home environment. Questions are answered using 4 points (1 = Very much like your own home, 4 = Non at all like your own home). Final scores are summed across the 15 items.
Lifestyle Behavior Checklist | Baseline
  Parent questionnaire: The Lifestyle Behavior Checklist is a 25 item, two-scale questionnaire. It is used to identify parental perception of problematic behaviors in the context of overweight and obesity (Problem Scale). The questionnaire also assesses the ability of the parent to deal with problematic behaviors (Confidence Scale). Each question on the Problem Scale is scored from 1 (not at all) to 7 (very much). Each question on the Confidence Scale is scored from 1 (Certain I can't do it) to 10 (Certain I can do i).
Binge Eating Scale | Baseline
  Parent questionnaire: The Binge Eating Scale (BES) is a 16-item questionnaire used to identify certain binge eating behaviors. < 17 indicates non-binging, 18-26 indicates moderate binging, and >27 indicates severe binging.
Family Food Behavior | Baseline
  Parent questionnaire: The Family Food Behavior Survey (FFBS) is a 20-item questionnaire that examines the degree to which adult monitor and make decisions about their child's eating behavior. Each of the 20 questions is scored using a 5 point Likert scale (0 = never true, 4 = always true). Their are four scales, (1). Maternal control of child feeding, (2). Maternal presence, (3). Child choice, (4). Organization. Higher scores on any scale indicate greater involvement by child or mother.
Sensitivity to Punishment and Reward | Baseline
  Parent questionnare: The Sensitivity to Punishment and Reward Questionnaire (SPSRQ) consists of 48 questions. Parents respond with "Yes" or "No" and it is scored on two scales. One scale is for sensitivity to punishment, and one scale is for sensitivity to reward. The items are summed to make a final score for each subscale.
Parent Weight Loss Behavior | Baseline
  Parent questionnaire: 24 item questionnaire assessing weight loss strategies over the last two years. Items are measured on a 5-point scale from 1 = Never, 5 = Always. There are 11 items relating to healthy weight loss factors and 9 items related to unhealthy weight loss factors.
Three Factor Eating | Baseline
  Parent Questionnaire: The Three Factor Eating Questionnaire - Revised 18 items - is an 18-item questionnaire assessing feelings and experiences towards eating behaviors. It is scored on three sub-scales: uncontrolled eating, cognitive restraint and emotional eating. Any items answered 1-2 are scored 1; 3-4 are scored as 2; 5-6 scored as 3, and 7-8 are scored as 4.
Parental Strategies to Teach about Advertising | Baseline
  Parent Questionnaire: The Parental Strategies to Teach about Advertising is a questionnaire assessing parental attitudes, beliefs and behaviors towards media and advertising use. There is no scaling used.
Structure and Control in Parent Feeding | Baseline
  Parent Questionnaire: The Structure and Control in Parent Feeding (SCPF) questionnaire assesses positive aspects of parental feeding practices. The Structure Model consists of 22 questions and the Control Model consists of 12 questions. The items are answered using a 5 points scale 0 = Never, 4 = Always.
Comprehensive Feeding Practices | Baseline
  Parent Questionnaire: The Comprehensive Feeding Practices Questionnaire is a 49-item, 12 factor survey. The factors include Monitoring, Emotional Regulation, Food as Reward. Child Control, Modeling, Restriction for Weight, Restriction for Health, Teaching Nutrition, Encourage Balance, Pressure to Eat, Healthy Environment and Involvement.
Comprehensive Feeding Practices | 1 Year
  Parent Questionnaire: The Comprehensive Feeding Practices Questionnaire is a 49-item, 12 factor survey. The factors include Monitoring, Emotional Regulation, Food as Reward. Child Control, Modeling, Restriction for Weight, Restriction for Health, Teaching Nutrition, Encourage Balance, Pressure to Eat, Healthy Environment and Involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Masterson TD, Stein WM, Beidler E, Bermudez M, English LK, Keller KL. Brain response to food brands correlates with increased intake from branded meals in children: an fMRI study. Brain Imaging Behav. 2019 Aug;13(4):1035-1048. doi: 10.1007/s11682-018-9919-8. PMID 29971684
- [Background] Kling SMR, Pearce AL, Reynolds ML, Garavan H, Geier CF, Rolls BJ, Rose EJ, Wilson SJ, Keller KL. Development and Pilot Testing of Standardized Food Images for Studying Eating Behaviors in Children. Front Psychol. 2020 Jul 21;11:1729. doi: 10.3389/fpsyg.2020.01729. eCollection 2020. PMID 32793062
- [Background] Masterson TD, Bermudez MA, Austen M, Lundquist E, Pearce AL, Bruce AS, Keller KL. Food commercials do not affect energy intake in a laboratory meal but do alter brain responses to visual food cues in children. Appetite. 2019 Jan 1;132:154-165. doi: 10.1016/j.appet.2018.10.010. Epub 2018 Oct 9. PMID 30312738
- [Background] English LK, Fearnbach SN, Lasschuijt M, Schlegel A, Anderson K, Harris S, Wilson SJ, Fisher JO, Savage JS, Rolls BJ, Keller KL. Brain regions implicated in inhibitory control and appetite regulation are activated in response to food portion size and energy density in children. Int J Obes (Lond). 2016 Oct;40(10):1515-1522. doi: 10.1038/ijo.2016.126. Epub 2016 Jul 26. PMID 27457416
- [Background] Keller KL, Kuilema LG, Lee N, Yoon J, Mascaro B, Combes AL, Deutsch B, Sorte K, Halford JC. The impact of food branding on children's eating behavior and obesity. Physiol Behav. 2012 Jun 6;106(3):379-86. doi: 10.1016/j.physbeh.2012.03.011. Epub 2012 Mar 16. PMID 22450261
- [Background] Fearnbach SN, English LK, Lasschuijt M, Wilson SJ, Savage JS, Fisher JO, Rolls BJ, Keller KL. Brain response to images of food varying in energy density is associated with body composition in 7- to 10-year-old children: Results of an exploratory study. Physiol Behav. 2016 Aug 1;162:3-9. doi: 10.1016/j.physbeh.2016.03.007. Epub 2016 Mar 10. PMID 26973134